CLINICAL TRIAL: NCT01081899
Title: The Effectiveness of the Liverpool Care Pathway in Improving End of Life Care for Dying Cancer Patients in Hospital. A Cluster Randomised Trial.
Brief Title: The Effectiveness of the LCP in Improving End of Life Care for Dying Cancer Patients in Hospital.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regional Palliative Care Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RFPS-2006-6-341619
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Cancer
Keywords: dying patients; cancer; hospital; Liverpool Care Pathways
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The LCP-I Program. (Experimental): The Italian version of the Liverpool Care Pathways version 11 for hospital) Programme.
  Interventions: Other: The LCP-I Program
- standard healthcare practices (No Intervention): No specific interventions are planned in the control wards.

INTERVENTIONS:
Other: The LCP-I Program — The LCP-I Program is a continuous quality Improvement Program of end-of-life care implemented by a Palliative Care Unit (PCU) in a hospital Medical Ward.
  Other Names: continuous quality Improvement Program
  Arms: The LCP-I Program.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the LCP-I Program in improving the quality of end-of-life care provided to cancer patients who die on hospital medical wards as compared to standard healthcare practices.

DETAILED DESCRIPTION:
The availability of an effective quality improvement program for the care of dying patients in hospitals is particularly relevant to the healthcare scenario. The LCP-I Program has provided enough evidence to justify a randomized trial to evaluate its effectiveness.

Although the core objective of the LCP-I is improving the quality of end of life care for dying patients, the Program targets the healthcare professionals working on the hospital ward. The only feasible method of assessing the effectiveness of this Program is by performing a cluster trial, where hospital wards are randomized to receive (or not to receive) the implementation of the LCP-I Program.

Pairs of eligible medical wards from different hospitals will be randomized to receive the experimental intervention (the LCP-I Program) or no intervention at all for the duration of the study.

The LCP-I Program will be implemented in the experimental ward by the PCU. The LCP-I Program has a duration of 6 months from the beginning of the intensive training. No intervention will be implemented in the control ward until the end of the evaluation.

Quality of end-of-life care will be evaluated for each pair of randomized wards for all eligible cancer deaths occurring in the six months after the conclusion of the LCP-I Program in the experimental ward.

ELIGIBILITY:
Ward level

Inclusion Criteria:

* "Medical", "General Medical" or "Internal Medical" ward;
* at least 25 cancer deaths on the ward per year;
* consent from the Hospital and Ward Management to participate to the trial;
* consent from an expert and skills-trained PCU to implement the LCP-I Program

Exclusion Criteria:

- in the hospital another Medical Ward has already been randomised.

Individual level

Inclusion Criteria:

- all cancer patients deceased in the ward during the evaluation period;

Exclusion Criteria:

- the deceased was a relative of a professional working in the hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Quality of end-of-life care provided to dying cancer patients and their families. | six months after the implementation of the LCP Program
  Measured through the Global Scale of the Italian version of the Toolkit "After-death Bereaved Family Member Interview" (Teno J, et al 2001).

SECONDARY OUTCOMES:
quality of communication between the healthcare professionals, patients and families | six months after the implementation of the LCP Program
  Measured through the specific Scales of the Italian version of the Toolkit "After-death Bereaved Family Member Interview" (Teno J, et al 2001).
quality of emotional support to family members before and after the patients' death | six months after the implementation of the LCP Program
  Measured through the specific Scales of the Italian version of the Toolkit "After-death Bereaved Family Member Interview" (Teno J, et al 2001).
coordination of care | six months after the implementation of the LCP Program
  Measured through the specific Scales of the Italian version of the Toolkit "After-death Bereaved Family Member Interview" (Teno J, et al 2001).
provision of care focusing on patient's individual needs | six months after the implementation of the LCP Program
  Measured through the specific Scales of the Italian version of the Toolkit "After-death Bereaved Family Member Interview" (Teno J, et al 2001).
patient's physical well-being through a better control of physical symptoms | six months after the implementation of the LCP Program
  Symptom scales (pain, breathlessness and vomiting) from the Italian version of VOICES (Costantini M, 2005)
quality of communication between hospital staff and GPs | six months after the implementation of the LCP Program
  interview with GPs
appropriateness of therapeutic and diagnostic procedures | six months after the implementation of the LCP Program
  Tool for recording all diagnostic and therapeutic procedures effectively performed during the last 3 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Costantini, MD, Principal Investigator — National Cancer Research Institute - Genoa (Italy)
Locations (1):
- National Cancer Research Institute, Genoa, Italy

REFERENCES:
- [Derived] Costantini M, Romoli V, Leo SD, Beccaro M, Bono L, Pilastri P, Miccinesi G, Valenti D, Peruselli C, Bulli F, Franceschini C, Grubich S, Brunelli C, Martini C, Pellegrini F, Higginson IJ; Liverpool Care Pathway Italian Cluster Trial Study Group. Liverpool Care Pathway for patients with cancer in hospital: a cluster randomised trial. Lancet. 2014 Jan 18;383(9913):226-37. doi: 10.1016/S0140-6736(13)61725-0. Epub 2013 Oct 16. PMID 24139708
- [Derived] Costantini M, Ottonelli S, Canavacci L, Pellegrini F, Beccaro M; LCP Randomised Italian Cluster Trial Study Group. The effectiveness of the Liverpool care pathway in improving end of life care for dying cancer patients in hospital. A cluster randomised trial. BMC Health Serv Res. 2011 Jan 24;11:13. doi: 10.1186/1472-6963-11-13. PMID 21261949